CLINICAL TRIAL: NCT00000477
Title: Cholesterol Reduction in Seniors Program (CRISP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 66; U01HL044315 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 1992-06

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypercholesterolemia; Myocardial Ischemia
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypercholesterolemia; Myocardial Ischemia | interventions — Lovastatin

INTERVENTIONS:
Drug: lovastatin

SUMMARY:
To conduct a pilot study to determine whether lowering elevated serum cholesterol levels with 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG CoA) reductase inhibitors reduced mortality due to the sequelae of atherosclerotic cardiovascular disease in older men and women.

DETAILED DESCRIPTION:
BACKGROUND:

Circulating levels of cholesterol, specifically cholesterol associated with the low-density lipoprotein (LDL) fraction, have been established by observational epidemiologic studies and by metabolic, pathologic, genetic studies in humans and selected animal models, and by randomized clinical trials as a major etiologic factor in coronary heart disease. The ratio between the percent reduction in coronary heart disease incidence and the percent reduction in cholesterol levels associated with treatment in randomized trials, approximately 2:1, is almost exactly that predicted by numerous observational epidemiologic studies of this relationship. However, the clinical trials demonstrating that lowering LDL-cholesterol levels reduces subsequent incidence of coronary heart disease events have been confined by and large to middle-aged men with hypercholesterolemia as in the Lipid Research Clinics Coronary Primary Prevention Trial (LRC-CPPT) or to men with established coronary heart disease as in the Coronary Drug Project (CDP). Experimental confirmation that cholesterol-lowering treatment is worthwhile after as well as before age 60 is lacking. Thus, although the guidelines issued in October 1987 by the National Cholesterol Education Program's (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults did not discriminate explicitly by age, the absence of direct evidence of efficacy led them to allow room for physician judgment in applying their recommendations to older patients. This uncertainty in the application of the NCEP guidelines to older men and women is a matter of considerable consequence to the public health.

Epidemiologic studies suggest that the prognostic power of cholesterol levels diminishes with advancing age. Subdivision of the participants in several cohort studies into those above or below age 50 at entry shows that the increment in coronary heart disease risk per increment in total or LDL cholesterol level is nearly always substantially lower in the older group. In the Framingham Heart Study, the study with the most follow-up data beyond age 60, a 0.5 percent increment in the coronary heart disease incidence rate was estimated per 1 mg/dl increment in plasma cholesterol level -- about 60 percent of the increment seen in middle-aged men and women. However, the absolute numbers of potentially preventable coronary heart disease deaths, 80 percent of which occur after age 65, and myocardial infarctions attributable to high plasma cholesterol levels in Framingham and other observational studies appear to increase with increasing age.

Previous clinical trials of cholesterol-lowering drugs have been weakened by their limited efficacy and acceptability to patients. In older patients, the administration of cholesterol-lowering drugs may be further complicated by interactions with drugs taken for other more pressing conditions. However, since the Food and Drug Administration approved the HMG CoA reductase inhibitor, lovastatin, in September 1987, the agent has been efficacious and well-tolerated by patients of all ages, and has been used increasingly widely.

In 1986, an ad hoc committee of the National Heart, Lung, and Blood Institute's Atherosclerosis, Hypertension, and Lipid Metabolism Advisory Committee (AHLMAC) recommended a randomized clinical trial of cholesterol-lowering using an HMG CoA reductase inhibitor in the elderly. The recommendation was endorsed by the full AHLMAC and approved by the National Heart, Lung, and Blood Advisory Council (NHLBAC) in May 1987. However, due to the high cost of such a trial and concerns about feasibility, an initiative for a two-year pilot study at five clinical centers was developed and approved by the NHLBAC in September 1988. The Request for Applications was released in February 1989 and awards made in July 1990.

DESIGN NARRATIVE:

There were five clinical centers and a coordinating center in the pilot study. There were four pre-randomization visits at four to six week intervals. Subjects were eligible for inclusion if their LDL cholesterol levels remained above 120 mg/dl after the introduction of the American Heart Association Step 1 Diet at Visit 2. Subjects were randomized to diet plus a low dosage of lovastatin (20 mg), diet plus a high dosage of lovastatin (40 mg), or to diet plus a placebo. End points were changes in blood lipid levels. Data on other blood chemistry values, as well as quality-of-life measures and coronary heart disease morbidity and mortality, were also collected. LDL cholesterol levels were measured at clinic visits six and twelve weeks after randomization and at twelve week intervals thereafter. Serum alanine aminotransferase levels were measured at six week intervals to determine liver function and slit lamp exams were performed before and after study medication to detect lenticular opacities. Subjects were followed for a minimum of six months and a maximum of fifteen months.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record

ELIGIBILITY:
Men and women, ages 65 and older, with elevated low-density lipoprotein cholesterol levels between 159 and 221 mg/dl at entry.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1990-07; Study Completion 1992-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Applegate — University of Tennessee; John Crouse — Bowman Gray School of Medicine; Donald Hunninghake — University of Minnesota; Robert Knopp — University of Washington; John LaRosa — George Washington University

REFERENCES:
- [Background] Stoy DB, Curtis RC, Dameworth KS, Dowdy AA, Hegland J, Levin JA, Sousoulas BG. The successful recruitment of elderly black subjects in a clinical trial: the CRISP experience. Cholesterol Reduction in Seniors Program. J Natl Med Assoc. 1995 Apr;87(4):280-7. PMID 7752281
- [Background] Davis CE, Applegate WB, Gordon DJ, Curtis RC, McCormick M. An empirical evaluation of the placebo run-in. Control Clin Trials. 1995 Feb;16(1):41-50. doi: 10.1016/0197-2456(94)00027-z. PMID 7743788
- [Background] LaRosa JC, Applegate W, Crouse JR 3rd, Hunninghake DB, Grimm R, Knopp R, Eckfeldt JH, Davis CE, Gordon DJ. Cholesterol lowering in the elderly. Results of the Cholesterol Reduction in Seniors Program (CRISP) pilot study. Arch Intern Med. 1994 Mar 14;154(5):529-39. doi: 10.1001/archinte.154.5.529. PMID 8122946
- [Background] Santanello NC, Barber BL, Applegate WB, Elam J, Curtis C, Hunninghake DB, Gordon DJ. Effect of pharmacologic lipid lowering on health-related quality of life in older persons: results from the Cholesterol Reduction in Seniors Program (CRISP) Pilot Study. J Am Geriatr Soc. 1997 Jan;45(1):8-14. doi: 10.1111/j.1532-5415.1997.tb00971.x. PMID 8994481